CLINICAL TRIAL: NCT04376983
Title: Effect of Implant-based Telerehabilitation in Patients With Heart Failure on Daily Physical Activity, Quality of Life and Exercise Capacity (TELE-RCT Study)
Brief Title: Effect of Implant-based Telerehabilitation
Acronym: TELE-CRT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, prof. dr. Paul Dendale, Prof. Dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TELE-CRT1
Record Dates: First submitted 2020-05-04; First posted 2020-05-06 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure; Telemedicine; Cardiac Resynchronisation Therapy
MeSH Terms: conditions — Heart Failure | interventions — Telerehabilitation

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients will get no intervention
- Intervention (Experimental): Patients will transmit their CRT data every week (first 6 weeks) and then every two week to the Heart Centre Hasselt. The physical activity data will be used to deliver a tailored motivational message to the patient to increase physical activity in this group.
  Interventions: Behavioral: Telerehabilitation for patients with a cardiac resynchronisation device

INTERVENTIONS:
Behavioral: Telerehabilitation for patients with a cardiac resynchronisation device — Using the device-measured physical activity to create tailored motivational messages and tips to the patients to increase physical activity
  Arms: Intervention

SUMMARY:
The TELE-RCT study is a prospective 2 arm randomized controlled trial recruiting patients with an implanted CRT device in Jessa Hospital Hasselt in Belgium.

DETAILED DESCRIPTION:
The TELE-RCT study is a prospective 2 arm randomized controlled trial recruiting patients with an implanted CRT device in Jessa Hospital Hasselt in Belgium. Subjects that do not violate any of the exclusion criteria and that have provided informed consent, will be asked to participate in the study. Patients that enter the study will be randomly assigned in a 1:1 ratio to the intervention or control group. Given the nature of the study, no blinding can be applied.

A cardiac resynchronization therapy (CRT) device is a battery operated device consisting of a pulse generator and thin, insulated wires called leads. The device sends electrical impulses throughout the heart to improve pump activity. This is particularly helpful in patients suffering from chronic heart failure, given that the pump activity in these patients is compromised.

Two types of CRT devices exist. On one hand a cardiac resynchronization therapy defibrillator (CRT-D), which functions as a normal pacemaker but can also sense arrythmias that can lead to sudden cardiac arrest. The device recognizes these arrhythmias and generates a defibrillation to stop the abnormal rhythm. On the other hand a cardiac resynchronization therapy pacemaker (CRT-P), which only functions as a pacemaker.

b. Study population

In order to be enrolled in the TELE-RCT study, subjects must meet all of the following inclusion criteria:

* Patients with an implanted CRT-D or CRT-P device in which monitoring of physical activity is possible
* CRT device must be implanted for at least three months
* Dutch speaking and understanding
* Evidence of a personally signed and dated informed consent, indicating that the subject (or a legally-recognized representative) has been informed of all pertinent aspects of the study
* Age ≥ 18 years
* CRT capable of transmitting data about physical activity in an interpretable manner
* Willingness and physically able to follow an email-based or SMS-based telemonitoring program and other study procedures in a 12 weeks follow-up period.
* Clinically stable without inducible ischemia or high-risk ventricular arrhythmia, confirmed by the last available maximal ergo-spirometry test
* Possession of smartphone or email address, which the patients regularly check, in order to receive feedback from the research staff

Subjects presenting with any of the following will not be included in the study:

* The presence of an absolute or relative contraindication to moderate- intensity exercise
* Participation in a cardiac revalidation program in the months before enrollment in the study
* Patients with planned interventional procedure or surgery in next three months
* Present cardiovascular complaints that might interfere with exertion: unstable angina, recent ICD shock etc.
* Participation in other cardiac rehabilitation program trials, focusing on exercise outcome
* Orthopedic, neurologic, or any other pathologic condition that makes the patient physically unable to follow an email-based or SMS-based telemonitoring program
* Any condition, which, in the opinion of the investigator, would make it unsafe or unsuitable for the patient to participate in this study or a life expectancy of less than three months based on investigator's judgment

  c. Recruitment All patients will be recruited from the department of Cardiology of Jessa Hospital Hasselt or during the consultations in Heart Center Hasselt. Patients who are eligible for participation will be contacted by the study staff to obtain further information. They will receive a brochure which explains the study on one of their appointments with their cardiologist.

Time schedule: First patient first visit (FPFV): 15th of November 2019 Last patient last visit (LPLV): 31st of December 2020 4. Study procedures

1. Patient information Eligible participants must sign informed consent prior to undergoing any study-specific procedures. They will be asked to read, understand and sign the informed consent form during the first meeting.

   At the start of the study, each patient enrolled in the trial will be assigned a unique identification number in order to ensure the anonymity. In addition, it enables the researchers to link all collected data (answers to questionnaires, test results etc.) to the right patient and thus combine the data to gain insight into the results.
2. Randomization The randomization in this study will be varied out with sealed envelopes to ensure concealed patient allocation. Patients will be randomized to either the intervention group (group A) or the control group (group B) in a 1:1 ratio. Patients in group A (intervention group) will receive the standard care for patients with chronic heart failure at the Jessa Hospital Hasselt, supplemented with regular feedback by email or SMS about their daily physical activity. Patients in group B (control group) will only receive the standard care for patients with chronic heart failure at the Jessa Hospital Hasselt.
3. Intervention Patients in the intervention group (group A) will receive standard care for patients with chronic heart failure and an implanted CRT device at Jessa Hospital Hasselt. The standard care consists of half-yearly appointments with a cardiologist and telemonitoring for arrhythmia. In addition to the standard care, the patients in the intervention group will also receive regular feedback about their physical activity. During the first 6 weeks of the trial, the patients in the intervention group will receive weekly feedback about their daily physical activity. During the following 6 weeks, patients will receive feedback every other week. The feedback will be given by study staff and will be sent to the patient by email or SMS. The type of feedback a patient will receive will be based on the minimum required daily physical activity for patients with chronic heart failure. By looking at previous data, the study staff will also try to motivate the patient to increase their daily physical activity. The patiënt's daily physical activity will be telemonitored using the internal accelerometer of their CRT device. They will be asked to manually transmit the data from their CRT device to the Jessa Hospital every week.

Patients in the control group (group B) will only receive the standard care Jessa Hospital Hasselt, being half-yearly appointments with a cardiologist and telemonitoring for arrhythmia.

ELIGIBILITY:
Inclusion Criteria:

* - Patients with an implanted CRT-D or CRT-P device in which monitoring of physical activity is possible
* CRT device must be implanted for at least three months
* Dutch speaking and understanding
* Evidence of a personally signed and dated informed consent, indicating that the subject (or a legally-recognized representative) has been informed of all pertinent aspects of the study
* Age ≥ 18 years
* CRT capable of transmitting data about physical activity in an interpretable manner
* Willingness and physically able to follow an email-based or SMS-based telemonitoring program and other study procedures in a 12 weeks follow-up period.
* Clinically stable without inducible ischemia or high-risk ventricular arrhythmia, confirmed by the last available maximal ergo-spirometry test
* Possession of smartphone or email address, which the patients regularly check, in order to receive feedback from the research staff

Exclusion Criteria:

* The presence of an absolute or relative contraindication to moderate- intensity exercise
* Participation in a cardiac revalidation program in the months before enrollment in the study
* Patients with planned interventional procedure or surgery in next three months
* Present cardiovascular complaints that might interfere with exertion: unstable angina, recent ICD shock etc.
* Participation in other cardiac rehabilitation program trials, focusing on exercise outcome
* Orthopedic, neurologic, or any other pathologic condition that makes the patient physically unable to follow an email-based or SMS-based telemonitoring program
* Any condition, which, in the opinion of the investigator, would make it unsafe or unsuitable for the patient to participate in this study or a life expectancy of less than three months based on investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Increase in percentage active minutes per day measured by CRT device | 12 weeks

SECONDARY OUTCOMES:
International Physical Activity Questionnaire | 12 weeks
HeartQol questionnaire | 12 weeks
Satisfaction: questionnaire | 12 weeks
SUS questionnaire | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Jessa Hospital, Hasselt, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No